CLINICAL TRIAL: NCT03212209
Title: A Crossover Study Comparing Fixed Continuous Airway Positive Pressure, FLEX- PLUS and Sensawake Modalities for OSA Treatment
Brief Title: Comparison of CPAP Modalities for OSA Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Fisher and Paykel Healthcare (Industry); Philips Respironics (Industry)
Responsible Party: Principal Investigator, Dalva Poyares, Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AssociacaoFIP
Record Dates: First submitted 2017-05-05; First posted 2017-07-11 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: This is a crossover study comparing different CPAP modalities in a group of patients with moderate to severe OSA.
Who Masked: Participant, Investigator
Masking Description: Participants have never had contact with CPAP, therefore were not aware of PAP modality prescribed. Investigator were also naive, as well as sleep specialist responsible for Polysomnography reports. Only respiratory therapist who was assigned to CPAP clinic was aware of patient´s treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- CPAP C- Flex-Plus by Philips Respironics (Experimental): Four consecutive weeks with CPAP C- FLEX PLUS treatment. After these 4 weeks, patients will undergo full PSG with CPAP FLEX- PLUS. Patients will also fill out Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, Functional Outcome Sleep Questionnaire, and visual analogue scale assessing CPAP side effects and patient´s comfort. Adherence to 4-week treatment will be checked. Treatment is followed by 7-day washout period.
  Interventions: Device: CPAP Fixed Pressure
- CPAP with Sensawake by Fisher and Paykel (Experimental): Four consecutive weeks with CPAP Sensawake treatment. After these 4 weeks, patients will undergo full PSG with the same CPAP modality. Patients will also fill out Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, Functional Outcome Sleep Questionnaire, and visual analogue scale assessing CPAP side effects and patient´s comfort. Adherence to 4-week treatment will be checked. Treatment is followed by 7-day washout period.
  Interventions: Device: CPAP Fixed Pressure
- CPAP fixed pressure (Active Comparator): Four consecutive weeks with CPAP fixed pressure treatment. After these 4 weeks, patients will undergo full PSG with the same CPAP modality. Patients will also fill out Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, Functional Outcome Sleep Questionnaire, and visual analogue scale assessing CPAP side effects and patient´s comfort. Adherence to 4-week treatment will be checked. Treatment is followed by 7-day washout period.
  Interventions: Device: CPAP Fixed Pressure

INTERVENTIONS:
Device: CPAP Fixed Pressure — Continuous positive airway pressure (CPAP) is the gold standard treatment for moderate and severe OSA, and it has been known to apply positive pressure in the upper airways, acting as a pneumatic splint preventing the upper airway collapse during sleep. CPAP C- Flex Plus by Philips - Respironics works just as CPAP Fixed Pressure, but increases the pressure delivered in the begining of inhalation to softens the breathing rhythm of the CPAP user. CPAP with SensAwake by Fisher and Paykel works just as CPAP fixed pressure but when the breathing pattern suggests that patient is awake, a prompt relief in pressure to the lowest most comfortable level is activated, like ramp feature.
  Other Names: CPAP C- Flex Plus by Philips Respironics; CPAP with SensAwake by Fisher and Paykel

SUMMARY:
This is a crossover study comparing the effect of CPAP Fixed Pressure, CPAP FLEX -PLUS and Sensawake on sleep quality, adherence to treatments, and PSG parameters in patients with moderate to severe OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is associated with behavioral, cognitive, metabolic and cardiovascular conditions. Continuous Positive Airway Pressure (CPAP) is the gold standard treatment for OSA. Despite being the most effective treatment for OSA, 46 to 83% of patients do not adhere to CPAP. New technologies for CPAP treatment have been developed in order to improve patient's comfort, adherence and effectiveness in reducing apnea, hypopneas and flow limitation events. As an example, the FLEX- PLUS technology which increases inspiratory positive pressure and decreases expiratory positive pressure would soften the rhythm of breathing. Sensawake is another technology which evaluates breathing pattern changes during CPAP therapy. When the breathing pattern suggests that patient is awake, a prompt relief in pressure is activated, like ramp feature. However, it is not clear whether CPAP FLEX- PLUS or Sensawake are superior compared with fixed pressure CPAP, in terms of polysomnographic parameters, especially flow limitation or adherence to treatment. Objective: To compare the effect of fixed pressure CPAP, CPAP FLEX- PLUS and Sensawake on sleep and compliance parameters in patients with moderate to severe OSA. Methods: Fifty male patients with moderate to severe OSA will be included in a crossover design study. All patients will use each CPAP modality for 30 days in a randomized order, namely CPAP with Fixed Pressure, Flex- PLUS and Sensawake. A week of washout period will be applied between treatments. All patients will wear the same nasal mask brand. At the end of each treatment (every 4 weeks), patients will undergo polysomnography and fill out Epworth, FOSQ, Pittsburgh questionnaires and a visual analogue scale assessing CPAP side effects and patient´s comfort. Finally, adherence to CPAP modalities will be systematically checked.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* apnea-hypopnea index (AHI) score of ≥20 events/hour of sleep
* 30-65 years-old
* body mass index (BMI) ≤40 Kg/m²

Exclusion Criteria:

* major neurological, psychiatric, cardiac or respiratory disease
* use of psychoactive medication
* other sleep disorders
* patients referred to PSG for Bilevel, considered the need for PAP ≥ 18 cm H2O
* Previous contact with any OSA treatment.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-02-14 (Estimated); Study Completion 2018-07-16 (Estimated)

PRIMARY OUTCOMES:
Flow limitation | 4 weeks after each CPAP modality completion
  Flow limitation in percentage of total sleep time. The flow limitation will be assessed by the flow curve obtained in the polysomnographic recording.

SECONDARY OUTCOMES:
Adherence to CPAP treatment | 4 weeks after each CPAP modality completion
  Adherence to CPAP treatment will be evaluated by CPAP SD card download data
Arousal index | 4 weeks after each CPAP modality completion
  Number of arousals per hour of sleep assessed by polysomnographic recording
Wake time after sleep onset | 4 weeks after each CPAP modality completion
  Wake time after sleep onset assessed by polysomnographic recording

CONTACTS AND LOCATIONS:
Overall Officials: Dalva Poyares, MD, PhD, Study Director — AFIP - Associação de fundo e incentivo a pesquisa
Locations (1):
- Evelyn Brasil, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
In case there is a future metanalysis in the subject, required by an indexed Journal or author.